CLINICAL TRIAL: NCT00347776
Title: Trial of Antibiotics to Reduce Recurrent Trichiasis (STAR)
Brief Title: Study of Azithromycin to Prevent Recurrent Trichiasis Following Surgery in Ethiopia
Acronym: STAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH); Project ORBIS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U01EY013878 (NIH)
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-06

CONDITIONS: Trichiasis
Keywords: trichiasis; azithromycin; trichiasis surgery; topical tetracycline
MeSH Terms: conditions — Trichiasis | interventions — Azithromycin; Tetracycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): topical tetracycline
  Interventions: Drug: topical tetracycline
- Intervention 1 (Active Comparator): oral azithromycin, single 1g dose to subject
  Interventions: Drug: azithromycin
- Intervention 2 (Active Comparator): single oral azithromycin dose to subject and immediate family members
  Interventions: Drug: azithromycin

INTERVENTIONS:
Drug: azithromycin — oral antibiotic
  Other Names: Zithromax
  Arms: Intervention 1; Intervention 2
Drug: topical tetracycline
  Arms: Control

SUMMARY:
Trachoma, an ocular infection caused by C. trachomatis, is the second leading cause of blindness worldwide.Years of repeated infection with C. trachomatis cause the eyelid to scar and contract and ultimately to rotate inward such that eyelashes rub against the eyeball and abrade the cornea (trichiasis). The World Health Organization (WHO) has endorsed a multi-faceted strategy to combat trachoma, which includes surgery to correct trichiasis. Despite this encouraging news, under the best of circumstances the recurrence rate of trichiasis following surgery is disappointingly high. The objective of our project is to conduct a randomized, controlled clinical trial of post-surgical antibiotic treatment, comparing oral azithromycin to topical tetracycline, for trichiasis surgical patients in Ethiopia with the goal of determining the impact of treatment on rates of trichiasis recurrence at one and two years.

DETAILED DESCRIPTION:
A randomized clinical trial of the effectiveness of a single dose of azithromycin compared to 6 weeks of topical tetracycline, and the added benefit of family-based azithromycin treatment, in preventing recurrence of trichiasis following surgery is proposed. This will provide the evidence base to inform and change the global public health policy and the donation program policy, regarding post-surgical treatment for trichiasis patients and possibly their families.

The investigators will determine the impact of three treatment strategies following trichiasis surgery on the rate of trichiasis recurrence in the operated eye at six months and one year. A randomized clinical trial of 1425 trichiasis surgical patients will be conducted in Sodo,Ethiopia. The first group (Control Group) will receive topical tetracycline following surgery; the second group (Intervention Patient Group) will receive oral azithromycin; the third group (Intervention Family Group) will receive oral azithromycin, and all family members resident in the patient's household will also receive oral azithromycin. Data will be collected at baseline (pre-surgery) on ocular status and infection status. Data will be collected at the time of surgery on surgery-related variables and surgical and post-operative complications. Additional data will be collected on any surgical complications and early recurrence at the two-week visit when sutures will be removed. A follow up visit at two months will include data collection on recurrence and presence of ocular infection. Evaluations for trichiasis recurrence will occur again at six months and at one year post-surgery. The latter visit will also include data collection on presence of ocular infection in the surgical case, and ocular infection in household members. Evaluation of the risk of recurrence at six months and one, two, and three years within each group will be completed to determine the benefit of using azithromycin compared to topical tetracycline, and the added benefit of family-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of trichiasis:
* no previous report of trichiasis surgery in at least one eye with trichiasis:
* Agreement by at least one other family member accompanying the patient that, if the patient is randomized to the family-treatment arm, s/he also would be willing to receive antibiotic treatment
* Age 18 or older

Exclusion Criteria:

* other household members concurrently participating in the trial
* Self-reported pregnancy
* Documented allergy to tetracycline
* Plans to move out of the region within 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1452 (Actual)
Dates: Start 2001-08; Primary Completion 2003-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila K West, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Melese M, West ES, Alemayehu W, Munoz B, Worku A, Gaydos CA, West SK. Characteristics of trichiasis patients presenting for surgery in rural Ethiopia. Br J Ophthalmol. 2005 Sep;89(9):1084-8. doi: 10.1136/bjo.2005.066076. PMID 16113353
- [Background] West ES, Munoz B, Imeru A, Alemayehu W, Melese M, West SK. The association between epilation and corneal opacity among eyes with trachomatous trichiasis. Br J Ophthalmol. 2006 Feb;90(2):171-4. doi: 10.1136/bjo.2005.075390. PMID 16424528
- [Background] West ES, Alemayehu W, Munoz B, Melese M, Imeru A, West SK. Surgery for Trichiasis, Antibiotics to prevent Recurrence (STAR) Clinical Trial methodology. Ophthalmic Epidemiol. 2005 Aug;12(4):279-86. doi: 10.1080/09286580591005769. PMID 16033749
- [Result] West SK, West ES, Alemayehu W, Melese M, Munoz B, Imeru A, Worku A, Gaydos C, Meinert CL, Quinn T. Single-dose azithromycin prevents trichiasis recurrence following surgery: randomized trial in Ethiopia. Arch Ophthalmol. 2006 Mar;124(3):309-14. doi: 10.1001/archopht.124.3.309. PMID 16534049
- [Derived] Woreta F, Munoz B, Gower E, Alemayehu W, West SK. Three-year outcomes of the surgery for trichiasis, antibiotics to prevent recurrence trial. Arch Ophthalmol. 2012 Apr;130(4):427-31. doi: 10.1001/archophthalmol.2011.374. Epub 2011 Dec 12. PMID 22159169
- [Derived] Gower EW, Merbs SL, Munoz BE, Kello AB, Alemayehu W, Imeru A, West SK. Rates and risk factors for unfavorable outcomes 6 weeks after trichiasis surgery. Invest Ophthalmol Vis Sci. 2011 Apr 25;52(5):2704-11. doi: 10.1167/iovs.10-5161. Print 2011 Apr. PMID 21051704
- [Derived] Woreta TA, Munoz BE, Gower EW, Alemayehu W, West SK. Effect of trichiasis surgery on visual acuity outcomes in Ethiopia. Arch Ophthalmol. 2009 Nov;127(11):1505-10. doi: 10.1001/archophthalmol.2009.278. PMID 19901217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomly assigned initially to receive single dose of oral azithromycin to subject or single dose of azithromycin to subject & immediate family members or topical tetracycline ointment to subject groups.1 yr data suggested no difference in outcome between 2 azithromycin arms.These 2 groups were combined into 1 group in final analysis.
Groups:
- Control: Topical tetracycline ointment to subject. Antibiotic: Topical tetracycline ointment administered twice daily for for 6 weeks
- Intervention 1: Oral azithromycin,single 1g dose to subject only Antibiotic : Oral azithromycin (1 g)
- Intervention 2: Oral azithromycin,single 1g dose to subject and immediate family members Antibiotic : Oral azithromycin (1 g)
Period: 1.5 Month Follow-up
Arm/Group | Control | Intervention 1 | Intervention 2
Started | 484 | 483 | 485
Completed | 470 | 475 (473 had no recurrence.2 were lost to follow-up but were still eligible for follow-up at next visits) | 473 (472 had no recurrence.1 was lost to follow-up but was still eligible for follow-up at next visits)
Not Completed | 14 | 8 | 12
Not completed — Death | 2 | 0 | 0
Not completed — reached the endpoint | 12 | 8 | 12
Period: 6 Month Follow-up
Arm/Group | Control | Intervention 1 | Intervention 2
Started | 470 | 475 | 473
Completed | 448 (440 had no recurrence.8 were lost to follow-up but were still eligible for follow-up at next visits) | 462 (459 had no recurrence.3 were lost to follow-up but were still eligible for follow-up at next visits) | 455 (452 had no recurrence.3 were lost to follow-up but were still eligible for follow-up at next visits)
Not Completed | 22 | 13 | 18
Not completed — Death | 2 | 1 | 3
Not completed — reached endpont | 20 | 12 | 15
Period: 12 Month Follow-up
Arm/Group | Control | Intervention 1 | Intervention 2
Started | 448 | 462 | 455
Completed | 425 | 446 | 436
Not Completed | 23 | 16 | 19
Not completed — Lost to Follow-up | 7 | 6 | 6
Not completed — Death | 3 | 4 | 4
Not completed — Reached endpoint | 13 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Intervention1: Oral azithromycin,single 1g dose to subject Antibiotic : Oral azithromycin (1 g)
- Intervention2: Oral azithromycin,single 1g dose to subject and immediate family members Antibiotic : Oral azithromycin (1 g)
- Total: Total of all reporting groups
Arm/Group | Control | Intervention1 | Intervention2 | Total
Number analyzed (Participants) | 484 | 483 | 485 | 1452
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (12.8) | 48.5 (13.0) | 50.0 (12.6) | 48.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 390 | 366 | 365 | 1121
  Male | 94 | 117 | 120 | 331
Region of Enrollment [Count of Participants; unit: Participants]
  Ethiopia | 484 | 483 | 485 | 1452

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Trichiasis in Tetracycline and Azithromycin Groups
Description: Recurrence of trichiasis : Clinical assessment was done by looking for one or more eye lashes touching globe or evidence of epilation.
Time Frame: Primary outcome assessed at 2 weeks,1.5 months, 6 months and 12 months post-surgery
Population: Recurrence rates (expressed as person-years) in the tetracycline arm was compared with the 2 azithromycin arms combined (483+ 485= 968 participants)
Measure: Count of Participants; unit: Participants
Groups:
- Control: Topical tetracycline
  Antibiotic:Topical tetracycline
- Intervention: The two azithromycin groups combined
  Antibiotic: Oral Azithromycin
Arm/Group | Control | Intervention
Number analyzed (Participants) | 484 | 968
Participants | 45 | 62
Statistical Analysis 1: Comparison: Control vs Intervention; The log rank test was done to compare the survival rates between the tetracycline arm and the azithromycin arms combined. The Cox proportional hazard model was used to evaluate risk factors and adjust for confounding in predicting recurrence; Test type: Superiority; p = .047, Log Rank; Cox Proportional Hazard = 0.67, 95% CI 2-sided [0.45 to 0.98]

2. Primary Outcome: Recurrent Trichiasis Between Two Azithromycin Arms
Description: Recurrence of trichiasis :Clinical assessment for recurrence was done by looking for one or more eye lashes touching globe or evidence of epilation.
  If there was evidence of epilation or if one or more eye lashes were touching the globe, it was considered as recurrence of trichiasis.
Time Frame: Primary outcome assessed at 2 weeks,1.5 months, 6 months and 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention1 | Intervention2
Number analyzed (Participants) | 483 | 485
Participants | 26 | 36
Statistical Analysis 1: Comparison: Intervention1 vs Intervention2; We tried to evaluate if treating the immediate family members of the subject with oral azithromycin along with the subject had added advantage in reducing the rate of recurrent trichiasis in comparison to treating the subject alone with oral azithromycin post surgery. The log rank test was done to compare the survival rates between the two intervention arms.The comparison results were expressed in person-years; Test type: Superiority; p = 0.19, Log Rank

3. Secondary Outcome: Surgical Failure
Description: The surgery was considered a failure if one or more eye lashes were touching the globe of the eye of the subject.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 484 | 968
Participants | 12 | 20
Statistical Analysis 1: Comparison: Control vs Intervention; Surgery was considered a failure if there was trichiasis recurrence at 6 week follow-up; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.36 to 1.10] — Comparison group was the tetracycline group

4. Secondary Outcome: Adverse Events
Description: At 6 weeks participants/family members were asked about any hospitalization,death,ocular complaints, gastrointestinal illness or other specific illness or any clinic visit within six weeks of receiving surgery.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 484 | 968
Participants
  Gastrointestinal complaints/other specific illness | 6 | 22
  Ocular complaints | 7 | 6

ADVERSE EVENTS:
Time Frame: At 1.5 months ( 6 weeks) post surgery.Adverse events were defined as death, hospitalization, gastrointestinal illness or other specific illness,ocular complaints. Events were assessed without regard to the specific Adverse Event Term.
Description: At the 1.5-month follow-up visit, specific questions were asked of each subject about himself/herself and all his/her family members about these adverse events.
  The interviewer was either a physician or a medical assistant
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 2/484 | 0/968
Serious Adverse Events (participants affected / at risk) | 0/484 | 0/968
Other Adverse Events (participants affected / at risk) | 13/484 | 28/968
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=484) | Intervention (N=968)
1.5 months (Surgical and medical procedures) | 6 | 22 — Gastrointestinal or other specific illness.Events were assessed without regard to the specific Adverse Event Term.At the 1.5-month follow-up,questions were asked from subject and all his/her family members about these adverse events.Adverse.
1.5 months (Surgical and medical procedures) | 7 | 6 — Ocular complaints. At the 1.5-month follow-up,questions were asked from subject and all his/her family members about these adverse events.Adverse Events were assessed without regard to the specific Adverse Event Term.

LIMITATIONS AND CAVEATS:
1.Azithromycin administered was observed.Compliance was 100%.In tetracycline group,only 1st application of ointment was observed.Data on compliance for next 6 weeks were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No